CLINICAL TRIAL: NCT04700150
Title: Effect of Tai Chi Protocol on Global Physical Activity in Patients With Spondyloarthitis in Comparison With a Control Group
Brief Title: Tai Chi in Spondyloarthritis
Acronym: TaiChiSpA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2018 SOUBRIER; 2018-A01275-50 (Other: 2018-A01275-50)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Spondyloarthritis
Keywords: SPONDYLOARTHITIS; TAI CHI CHUAN; PHYSICAL ACTIVITY
MeSH Terms: conditions — Spondylarthritis; Motor Activity | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group A (Experimental): 2 tai chi session per week during 4 month (M0 to M4)
  Interventions: Other: Tai Chi 4 month
- Control group B (Placebo Comparator): 2 tai chi session per week during 2 month (M2 to M4)
  Interventions: Other: Tai Chi 2 month

INTERVENTIONS:
Other: Tai Chi 2 month — Tai chi sessions will consist of repetition of simple and basic movements focusing mainly on breathing, relaxation and body diagram. This Chinese martial art also includes coordination exercises of body parts (legs, arms, pelvis and spine), looseness and limbering up of joints and muscles.
  Arms: Control group B
Other: Tai Chi 4 month — Tai chi sessions will consist of repetition of simple and basic movements focusing mainly on breathing, relaxation and body diagram. This Chinese martial art also includes coordination exercises of body parts (legs, arms, pelvis and spine), looseness and limbering up of joints and muscles.
  Arms: interventional group A

SUMMARY:
Our hypothesis is that tai chi sessions would increase physical activity of patients with Spondyloarthitis. The main objective is to study the effect of tai chi sessions (16 vs.0) on global physical activity of Spondyloarthitis patients, compared to a control group without tai chi.

DETAILED DESCRIPTION:
Selection and inclusion of patients will be done by principal investigator of Rheumatology Department. After verification of inclusion and non-inclusion criteria by principal investigator and signature of consent, patients will be randomized by 1: 1 randomization (centralized randomization by statistician into 2 groups at M0). They will participate in sessions in a deferred manner due to two per week for each group:

* Interventional "A" group: 32 sessions (on average 2/week) performed from M0 to M4 in 15 patients.
* Control "B" group: 16 sessions (on average 2/week) performed from M2 to M4 in 15 patients.

Patients of "B" group will be not performing sessions with "A" group patients. Sessions lasting about 45 minutes will be proposed from Monday to Friday in a room planned from this activity within the CHU. Exercises will be adapted and personalized according to each one. Evaluations will be carried out at M0, M2 and at the end of the protocol at M4.

Assessment of pain and stress will be done before and after each session. Final assessment will be done at 4 months after randomization. Fitness assessment and tai chi sessions will be conducted by APA student.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old with Spondyloarthitis (ASAS criteria), with activity deemed stable by rheumatologist.
* Patient able to walk without help
* Patient able to complete a questionnaire
* Patient giving informed consent.
* Patient covered by social security

Exclusion Criteria:

* Patient with disorder of higher mental function or psychiatric disorders.
* Patient who has previously contribute to a tai chi program.
* Patient with an absolute contraindication to physical activity.
* Protected populations: pregnant women, breastfeeding women, tutorship, trusteeship, deprived of liberty, safeguard of justice

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Change in global physical activity time per week, Global Physical Activity Questionnaire | Month 0
  measured by modified Global Physical Activity Questionnaire (GPAQ) .
Change in global physical activity time per week, Global Physical Activity Questionnaire | Month 2
  measured by modified Global Physical Activity Questionnaire (GPAQ) .
Change in global physical activity time per week, measured by an accelerometer | Month 0
  measured by an accelerometer between M0 and M2 expressed in MET.min/week.
Change in global physical activity time per week, measured by an accelerometer | Month 2
  measured by an accelerometer between M0 and M2 expressed in MET.min/week.

SECONDARY OUTCOMES:
Change in Physical activity time of light intensity, moderate intensity, high intensity | Month 0
  measured by an accelerometer
Change in Physical activity time of light intensity, moderate intensity, high intensity | Month 2
  measured by an accelerometer
Change in Physical activity time of light intensity, moderate intensity, high intensity | Month 4
  measured by an accelerometer
Change in Physical activity time of light intensity, moderate intensity, high intensity | Month 0
  measured by the modified Global Physical Activity Questionnaire
Change in Physical activity time of light intensity, moderate intensity, high intensity | Month 2
  measured by the modified Global Physical Activity Questionnaire
Change in Physical activity time of light intensity, moderate intensity, high intensity | Month 4
  measured by the modified Global Physical Activity Questionnaire
Change in Sedentary time | Month 2
  measured by modified Global Physical Activity Questionnaire
Change in Sedentary time | Month 4
  measured by modified Global Physical Activity Questionnaire
Change in Sedentary time | Month 2
  measured by an accelerometer
Change in Sedentary time | Month 4
  measured by an accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soubrier, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Fayet F, Fan A, Pereira B, Lambert C, Perron L, Rodere M, Duclos M, Soubrier M. Effects of face-to-face and remote Tai Chi in stable axial spondyloarthritis: a pilot randomised controlled trial. Rheumatol Int. 2025 Aug 1;45(8):178. doi: 10.1007/s00296-025-05912-5. PMID 40748484